CLINICAL TRIAL: NCT04263337
Title: Neurologic Function Across the Lifespan: A Prospective, LONGitudinal, and Translational Study for Former National Football League Players
Brief Title: NFL LONG Prospective Study
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Boston Children's Hospital (Other); Medical College of Wisconsin (Other); National Football League (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 19-1065
Record Dates: First submitted 2020-01-31; First posted 2020-02-10 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Concussion, Brain
Keywords: Concussion; Former NFL Players; Football; Neurologic; Sub-concussive Exposure
MeSH Terms: conditions — Brain Concussion; Neurologic Manifestations | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole; 2-(6-chloro-2-(4-(3-fluoropropoxy)phenyl)imidazo(1,2-a)pyridin-3-yl)-N,N-diethylacetamide; 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Low Cognitive Functioning/Low Concussion History (Other): Former NFL players with low cognitive function and low concussion history will be included in this group.
  Interventions: Drug: [11C] PiB; Drug: [18F] PBR111; Drug: [18F] Flortaucipir
- High Cognitive Functioning/ High Concussion History (Other): Former NFL players with high cognitive function and high concussion history will be included in this group.
  Interventions: Drug: [11C] PiB; Drug: [18F] PBR111; Drug: [18F] Flortaucipir
- Low Cognitive Functioning/High Concussion History (Other): Former NFL players with low cognitive function and high concussion history will be included in this group.
  Interventions: Drug: [11C] PiB; Drug: [18F] PBR111; Drug: [18F] Flortaucipir
- High Cognitive Functioning/Low Concussion History (Other): Former NFL players with high cognitive function and low concussion history will be included in this group.
  Interventions: Drug: [11C] PiB; Drug: [18F] PBR111; Drug: [18F] Flortaucipir
- Healthy Male Controls (Other): Healthy male demographically matched controls will be included in this group.
  Interventions: Drug: [11C] PiB; Drug: [18F] PBR111; Drug: [18F] Flortaucipir
- Low Cognitive Functioning/Medium Concussion History (Other): Former NFL players with low cognitive function and medium concussion history will be included in this group.
  Interventions: Drug: [11C] PiB; Drug: [18F] PBR111; Drug: [18F] Flortaucipir
- Medium Cognitive Functioning/Low Concussion History (Other): Former NFL Players with medium cognitive functioning and low concussion history with be included in this group.
  Interventions: Drug: [11C] PiB; Drug: [18F] PBR111; Drug: [18F] Flortaucipir
- Medium Cognitive Functioning/Medium Concussion History (Other): Former NFL Players with medium cognitive functioning and medium concussion history with be included in this group.
  Interventions: Drug: [11C] PiB; Drug: [18F] PBR111; Drug: [18F] Flortaucipir
- Medium Cognitive Functioning/High Concussion History (Other): Former NFL Players with medium cognitive functioning and high concussion history with be included in this group.
  Interventions: Drug: [11C] PiB; Drug: [18F] PBR111; Drug: [18F] Flortaucipir
- High Cognitive Functioning/Medium Concussion History (Other): Former NFL Players with high cognitive functioning and high concussion history with be included in this group.
  Interventions: Drug: [11C] PiB; Drug: [18F] PBR111; Drug: [18F] Flortaucipir

INTERVENTIONS:
Drug: [11C] PiB — Per study protocol static PET images will be acquired after IV infusion of CPiB to generate standard uptake values (SUVs). PET imaging is necessary in order to address the primary and secondary outcome measures as a component of neurological health (i.e., presence of proteinopathies empirically associated with neurodegenerative disease, cognitive decline, and neurological signs/symptoms). All groups will participate in this portion of the protocol.
  Other Names: C11 PiB Amyloid
Drug: [18F] PBR111 — Per study protocol static PET images will be acquired after IV infusion of F-PBR111 to generate standard uptake values (SUVs). PET imaging is necessary in order to address the primary and secondary outcome measures as a component of neurological health (i.e., presence of proteinopathies empirically associated with neurodegenerative disease, cognitive decline, and neurological signs/symptoms). All groups will participate in this portion of the protocol.
  Other Names: F18 PBR-111
Drug: [18F] Flortaucipir — Per study protocol static PET images will be acquired after IV infusion of F-T807 to generate standard uptake values (SUVs). PET imaging is necessary in order to address the primary and secondary outcome measures as a component of neurological health (i.e., presence of proteinopathies empirically associated with neurodegenerative disease, cognitive decline, and neurological signs/symptoms). All groups will participate in this portion of the protocol.
  Other Names: F18 T807 Tau

SUMMARY:
The purpose of this 5-year prospective research study is to characterize the association between concussions, sub-concussive exposure, and long-term neurologic health outcomes in former NFL players. To achieve the study aims, the investigators will conduct detailed research visits that include clinical outcome assessments, blood-based biomarkers, advanced magnetic resonance imaging (MRI), positron emission tomography (PET) using investigational tracers and genetic testing. Ultimately, the goal of this study is to translate the findings from this study into clinical, interventional studies for at risk former NFL players.

DETAILED DESCRIPTION:
There is growing concern that repetitive concussions, or even exposure to sub-concussive blows during collision sports, may be associated with chronic neurologic problems, including CTE. Despite the lay media attributing devastating clinical problems to CTE, no studies conclusively demonstrate a connection between the pathological findings and clinical effects. Experts at the 5th International Conference on Concussion concluded that "a cause-and-effect relationship has not yet been demonstrated between CTE and SRCs [sport-related concussions]" and "the notion that repeated concussion or sub-concussive impacts cause CTE remains unknown." As there are no treatments or prevention strategies available for CTE, some former players who attribute their problems to CTE develop depression, despair, and suicidality. There is a pressing need to understand the risk, incidence, character, progression, and treatment of the neurologic health problems of former NFL players.

The investigators propose an in-depth study assessing the association between concussion, sub-concussive exposure, cerebral tau, and clinical outcomes; assessing former NFL players for autoantibodies to cis-tau; assessing carbon monoxide (CO), memantine, environmental enrichment (EE), and cis P-tau antibodies for preventing and treating neurologic sequela of rmTBI. The most promising treatment(s) from preclinical studies will ultimately be translated into clinical trials for individuals identified during the clinical study who are at risk for long-term neurologic health problems. The study will be carried out at 2 sites, The University of North Carolina at Chapel Hill and The Medical College of Wisconsin both at the oversight of the main grant awardee, Boston Children's Hospital.

In order to prospectively and longitudinally track progression of neurologic health and assess associations with concussion and sub-concussive exposure the investigators plan to execute multiple study phases: (1) Former National Football League (NFL) Players will complete the General Health Survey (GHS)(part of a previous research study); (2) Stratification based on age and the GHS; (3) Phone Screening with Brief Test of Adult Cognition by Telephone (BTACT); (4) Re-stratification based on BTACT scores; (5) In-Person Neurobiopsychosocial Research Evaluation 1; (6) Annual Follow-Up Health Surveys; and (7) In-Person Neurobiopsychosocial Research Evaluation 2.

Based on the stratification above, 250 subjects will be enrolled for In-Person Research Evaluation 1. This cohort will include 100 high cognitive functioning former NFL players, 100 low cognitive functioning former NFL players, and a group of 50 demographically matched healthy controls. Informants of the former NFL subjects, that are selected for In-Person Research Evaluation 1, will also be asked to complete a series of informant-based questionnaires (n=200). Subjects enrolled in the In-Person Research Evaluation 1 will complete an assessment of neurobiopsychosocial function, to include a detailed neuropsychological assessment, patient-reported outcomes, and symptom validity measures. Assessment of neurobiopsychosocial function will also include proteomic and genomic studies, multi-modal magnetic resonance imaging (MRI) and position emission tomography (PET) molecular imaging studies of tau, amyloid and inflammation.

Annual follow-up surveys of health status and life function (selected repeat measures from the GHS) will be sent/administered annually for 5 years. Based upon the annual follow-up survey of health status and life function, a subset of former NFL players and all controls will return for second a research assessment of neurobiopsychosocial function that mirrors the in-person research evaluation.

ELIGIBILITY:
Inclusion Criteria for Former NFL Player Group:

* At least 1 year of participation in National Football League (NFL groups)
* Retired from professional football
* Ages between 50-70

Inclusion Criteria for Healthy Controls:

* No prior exposure to football, collision sports, or prior concussions
* They will be matched to former NFL players by age and estimated premorbid intellectual functioning.
* Ages between 50-70

Exclusion Criteria:

* Any contraindications to MRI, PET, or biological study procedures
* History of Moderate or Severe TBI
* Current primary Axis I diagnosis of Psychotic Disorder
* History or clinical suspicion of other conditions (e.g., epilepsy, stroke, dementia) known to cause cognitive dysfunction
* Diagnosis /associated treatment that would preclude participation in full study protocol (e.g., terminal cancer)

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
PET Neuroimaging SUVR Over Time | Baseline, up to 3 Year Follow-up
  Positron Emission Tomography (PET) Scan- Standard uptake value ratio (SUVR) of the following tracers: Tau tracer, [18 F]Flortaucipir; AV1415 Amyloid tracer, Pittsburgh compound-B (11C-PiB); Neuroinflammation tracer, [18 F] peripheral benzodiazepine receptor (PBR111)
MRI Neuroimaging Over Time | Baseline, up to 3 Year Follow-up
  Advanced MRI Sequence Structural imaging (T1, T2, T2-FLAIR) Tissue/microstructural organization-Diffusion MRI Cerebral blood flow-Arterial Spin Labeling Susceptibility weighted imaging/quantitative susceptibility mapping Functional MRI- resting state functional MRI
Serum Biomarkers Over Time | Baseline, up to 3 Year Follow-up
  Blood collection for analysis of serum markers of neurodegenerative disease and neurodegeneration
Mean Change in Headache Impact Test (HIT-6) | Baseline, up to 3 Year Follow-up
  The HIT-6 is a screening measure that assesses the degree to which individual's experiences of headaches impacts their ability to perform daily functional roles. The six-items can be responded to in five ways, which include, never (6-points), rarely (8-points), sometimes (10-points), very often (11-points), and always (13-points).
Mean Change in MDS-UPDRS Score | Baseline, up to 3 Year Follow-up
  The MDS-UPDRS evaluates motor and non-motor symptoms in persons with Parkinson's and consists of 4 parts with various questions and evaluations. Parts I and II (non-motor) each contain 13 questions/evaluations, Part III (motor) contains 33 and Part IV (motor) contains 6. Each question/evaluation score ranges from 0 (normal) to 4 (severe). Higher scores indicate a greater impact of Parkinson's disease symptoms (i.e., worse symptoms).
Mean Change in Postural Stability-Sensory Organization Test | Baseline, up to 3 Year Follow-up
  The stability-sensory organization test is an index obtained by the NeuroCom Balance System. The minimum score is 0 and there is no specified maximum value. A lower score indicates better postural stability. Postural stability is measured utilizing a dynamic force plate to quantify the vertical forces exerted through the patient's feet to measure center of gravity position and postural control.
Mean Change in Structured Inventory of Malingered Symptomatology (SIMS) | Baseline, up to 3 Year Follow-up
  A 75 true-or-false item measures that assesses malingering psychopathology and neuropsychological symptoms. The measure provides an overall score for probably malingering, as well as five subscales; including Psychosis, Low Intelligence, Neurologic Impairment, Affective Disorders, and Amnestic Disorders Endorsement of highly atypical symptoms and endorsement pattern profiles, this measure has demonstrated efficacy in differentiating malingerers from true clinical populations.
Mean Change in Medical Symptom Validity Test (MSVT) | Baseline, up to 3 Year Follow-up
  The MSVT is measure typically used in the detection of suboptimal effort. The test consists of a process in which participants are asked to learn 10 word pairs and later recall the word pairs. The minimum score is 0% and the maximum value is 100%.
Mean Change in National Institute of Health (NIH) Toolbox | Baseline, up to 3 Year Follow-up
  A computerized measure of cognitive functioning across several domains of cognition developed by the NIH. The Toolbox Cognition measure is comprised of several subtests assessing various domains of cognitive functioning. The minimum score is 0 and there is no maximum score.
Mean Change in Rey Auditory Verbal Learning Test (RAVLT) | Baseline, up to 3 Year Follow-up
  The RAVLT is a measure of auditory verbal learning, which is commonly affected among individuals with memory and other related cognitive disorders. Subjects are asked the learn and immediately recall a 15-word list across 5 different trials. They are asked to do the same for second, intrusion list, and then they are asked to recall the first list immediately after. Following a 30 minute delay, participants are asked to spontaneously recall the word list. Immediately following the delay recall trial, recognition memory is tested in a yes/no format where subjects are asked to discriminate words from the original list from novel distractors. The minimum score is 0 and the maximum score is 15.
Mean Change in Dot Counting Test | Baseline, up to 3 Year Follow-up
  The Dot Counting Test is a measure effort and validity of session results. Within the measure, subjects are essentially asked to count the number of dots on various stimuli pages. Each specific page has a maximum ranging from 7-28 and the minimum score is 0.
Mean Change in Delis Kaplan Executive Function System (DKEFS) Verbal Fluency, Trailmaking Test (TMT), and Color-Word Interference | Baseline, up to 3 Year Follow-up
  The DKEFS is a measure that is associated with integrity and functioning of the frontal system of the brain, or executive functioning. Verbal fluency involves administration of 3 trials in which participants generate words based on letter prompts. The minimum score is 0 and there is no maximum. Two additional trials involving generation of word lists based on categories is also included. The DKEFS TMT is a test of speeded sequencing and set-shifting with sensitivity to sport-related concussion. There are 4 trials consisting of psychomotor speed, number sequencing, letter sequencing, and letter-number sequencing/shifting. The minimum is 0 and there is no maximum. DKEFS Color-Word consists of 4 trials in which participants are timed on (1) colors on the page, (2) read words on the page, (3) inhibit responses of words and state colors that items are printed in, and (4) set-shift in their ability to perform number 3 based on different principles. The minimum is 0 and there is no maximum.
Mean Change in Satisfaction with Life Scale (SWLS) Score | Baseline, up to 3 Year Follow-up
  Satisfaction with Life Scale is a short 5-item instrument designed to measure global cognitive judgments of satisfaction with one's life. Questions are responded to on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Total scores can be classified at extremely satisfied (31-35), satisfied (26-30), slightly satisfied (21-25), neutral (20), slightly dissatisfied (15-19), dissatisfied (10-14), and extremely dissatisfied (5-9).
Mean Change in Alcohol Use Disorders Identification Test (AUDIT) score | Baseline, up to 3 Year Follow-up
  Alcohol Use Disorders Identification Test consists of three domains: Hazardous alcohol use (items 1-3), dependence symptoms (items 4-6), and harmful alcohol use (items 7-10). Participants respond to items on a scale between 0 to 4, and a total score can be calculated based on individual items.
Mean Change in PROMIS Cognitive Functioning Score | Baseline, up to 3 Year Follow-up
  The PROMIS Cognitive Function is a self-reported measure that assesses patient-perceived cognitive deficits and the extent to which cognitive impairments interfere with daily functioning. The short-form consists of 4-itens that are scored on a 5-point Likert scale (5-never) to 1 (very often). Raw scores are converted into T-score for each participant. A T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Mean Change in WAIS-IV Coding and Symbol Search | Baseline, up to 3 Year Follow-up
  The Coding and Symbol Search subtests of the Wechsler Adult Intelligence Scale-Fourth Edition (WAIS-IV) are two subtests that make up the Processing Speed Index of the WAIS-IV. Each subtest requires two minutes to complete and ultimately, reflect the participants ability to complete as many items correctly as possible within the time limit. The minimum score is 0 and the maximum is 60 for Symbol Search and 135 for Coding.
Mean Change in Neuro-Quality Of Life (QOL): Emotional and Behavioral Dyscontrol | Baseline, up to 3 Year Follow-up
  This is an eight-item measure from the Neuro-QOL set of tools, which assesses various symptoms and behaviors associated with frontal lobe dysfunction, particularly as it relates to disinhibited actions or behaviors. Items are scored on a five-point Likert scale, ranging from 1 (never) to 5 (always). A T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Mean Change in Frontal systems behavior scale (FrsBe) | Baseline, up to 3 Year Follow-up
  The FrSBe is a 46-item self-report measure of various symptoms and behaviors commonly associated with executive dysfunction. On a 5-point Likert scale ranging from 1 to 5, participants endorse the degree to which they experience the symptom/behavior before and after the present illness/injury. A total frontal systems score can be calculated for before and after the injury/illness, as well as three subscales of frontal lobe symptoms or behaviors, including apathy, disinhibition, and executive dysfunction. Raw scores are converted into T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Mean Change in Everyday Cognition assessment (ECog) | Baseline, up to 3 Year Follow-up
  This measure is intended to be used as a measure of behaviors typically associated with forgetfulness and other cognitive difficulties. This will aid in identifying neurological health difficulties (i.e., cognitive decline) among those individuals who have limited insight on self-report cognitive functioning measures. The ECog Assessment is comprised of 12-items that are rated on a 4-point Likert scale ranging from 1 (better or no change compared to 10 years earlier) to 4 (consistently much worse). Total scores from the measure are calculated by summing responses on all items and dividing by the number of questions answered.
Mean Change in Minnesota Multiphasic Personality Inventory (MMPI)-2-RF Cognitive Complaints Scale | Baseline, up to 3 Year Follow-up
  The cognitive complaints scale is a subscale of the derived from the full MMPI-2-RF. As part of the full instrument, the Cognitive Complaints Scale has been used as an embedded measure of symptom validity. In order to avoid administering the full over 500 item instrument, only the 13-itmes from the Cognitive Complaints Scale are administered in isolation for the current study. Items are presented in a true-false format. This method of administration has been performed in a number of studies in the published literature. A T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Mean Change in PROMIS_29 Score | Baseline, up to 3 Year Follow-up
  A self-report 29-itme measure of overall functioning. Participants respond on a Likert scale ranging from 5 (without any difficulty) to 1 (unable to do). The measure generates an overall score of functioning, as well as subscales of physical function, anxiety, depression, fatigue, sleep disturbance, able to participate in social roles/activities, pain interference, and pain intensity. Raw scores are converted into T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Mean Change in Beck Depression Inventory (BDI-II) Score | Baseline, up to 3 Year Follow-up
  A 21-item measure inquiring about common symptoms of depression. Each item is measured on a scale from 0-3, with higher numbers reflecting a higher-degree of symptomology over the last 2 weeks for that item. Raw scores can be classified into severity categories, including normal (0-13), mild (14-19), moderate (20-28), and severe (29-63).
Mean Change in Beck Anxiety Inventory (BAI-II)-Score | Baseline, up to 3 Year Follow-up
  A 21-item measure of common physiological and worry-related symptoms associated with anxiety. Responses are recorded on a 4-point Likert scale ranging from 0 (not at all) to 3 (severely). Raw scores can be classified into severity categories, including minimal anxiety (0-7), mild anxiety (8-15), moderate (16-25), and severe (26-63).
Mean Change in Neuropsychiatric Inventory Questionnaire NPI-Q2 Score | Baseline, up to 3 Year Follow-up
  A measure of common dementia-related behavioral symptoms among older adults. Within the measure 12 domains of these symptoms are recorded, including delusions, hallucinations, agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, irritability/lability, and aberrant motor activity night-time behavioral disturbances and appetite, and eating abnormalities. A screening question is asked about each sub-domain. If the responses to these questions indicate that the patient has problems with a particular sub-domain of behavior, the caregiver is only then asked all the questions about that domain, rating the frequency of the symptoms on a 4-point scale, their severity on a 3-point scale, and the distress the symptom causes them on a 5-point scale.
Mean Change in Social Readjustment Rating Scale (SRRS) Score | Baseline, up to 3 Year Follow-up
  This 43-item measure quantifies stress associated with common life events (life changing unit), with a unique value associated with each event over a 12-month period. For example, death of a spouse garners a score of 100 and major holidays equals 11 points. The total number of points is summed and a higher score is representative of a greater degree of life-event related distress. A score of 150 life units or less suggests a 30% change of suffering from stress, 150-299 is associated with a 50% chance of suffering from stress, and over 300 life units suggests that the person has an 8% chance of developing a stress related illness.
Mean Change in Ego Resilience Scale (ER89) Score | Baseline, up to 3 Year Follow-up
  This is a 14-item measure used to assess resilience in individuals following stressful events. Items are scored on a 4 point Likert Scale ranging from 1-Does not Apply at All, 2-Applies Slightly, 3-Applies Somewhat, and 4- Applies Very Strongly; and scores for each item are summed to obtain a total score. Higher scores indicate a more favorable outcome
Mean Change in Athlete Identity Questionnaire Score | Baseline, up to 3 Year Follow-up
  This questionnaire has been adapted from the previously established "Athletic Identity Measurement Scale" for currently active athletes (not retired). Items are scored on a 7 point Likert Scale ranging from 1-Strongly Disagree to 7-Strongly Agree.
Mean Change in Childhood Development and Adversity Questions Score | Baseline, up to 3 Year Follow-up
  This is a 33-item questionnaire that was developed from previous work to give insight into childhood experiences, socioeconomic stability, and other important environmental factors that may influence later-life socioeconomic factors, health, and well-being. The questionnaire contains items pertaining to Social and Community Context (1 item), Economic Stability (4 items), Education Access and Quality (1 item), Health Care Access and Quality (2 items), Neighborhood and Built Environment (3 items), and Adverse Childhood Experiences (Emotional Neglect [6 items], Financial Need [2 items], Parental Intimidation [4 items], Parental Violence [2 items], and Family Problems and Separation [4 items]).
Mean Change in International Physical Activity Questionnaire (IPAQ) Score | Baseline, up to 3 Year Follow-up
  This is a 4-item questionnaire intended to obtain data on health-related physical activity. It was developed for both research studies and patient monitoring. Each of the 4 items asks about the number of days per week, and the duration of time in each day participating in different physical activities: vigorous; moderate; walking; and sitting. Answers to these questions will be used to compare to activity recommendations put forth by organizations such as the American College of Sports Medicine.
Mean Change in Rapid Eating Assessment for Participants (REAPS) Score | Baseline, up to 3 Year Follow-up
  This is a 16-item questionnaire about the individuals' behaviors regarding food consumption. Participants respond to the first 13 items by selecting from the following options: "Usually/often"; "Sometimes"; "Rarely/Never"; or, when appropriate, a selection that the item does not apply to them. Responses from these first 13 items are then scored and summed into a diet quality score, where the total range of values falls between "13" (lowest quality diet) and "39" (highest quality diet). Items 14 and 15 request "Yes" or "No" responses: 14. "You or a member of your family usually shops and cooks rather than eating sit-down or take-out restaurant food?"; and 15. "Usually feel well enough to shop or cook." The 16th item is answered on a 5-point Likert scale from "1" (Very willing) to "5" (Not at all willing).

CONTACTS AND LOCATIONS:
Overall Officials: William Meehan, MD, Principal Investigator — Boston Children's Hospital; Michael McCrea, PhD, Principal Investigator — Medical College of Wisconsin; Jason Mihalik, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- United States (3):
  - Boston Children's Hospital, Waltham, Massachusetts
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Randolph C, Karantzoulis S, Guskiewicz K. Prevalence and characterization of mild cognitive impairment in retired national football league players. J Int Neuropsychol Soc. 2013 Sep;19(8):873-80. doi: 10.1017/S1355617713000805. Epub 2013 Aug 1. PMID 23902607
- [Background] Guskiewicz KM, Marshall SW, Bailes J, McCrea M, Cantu RC, Randolph C, Jordan BD. Association between recurrent concussion and late-life cognitive impairment in retired professional football players. Neurosurgery. 2005 Oct;57(4):719-26; discussion 719-26. doi: 10.1093/neurosurgery/57.4.719. PMID 16239884
- [Background] Kerr ZY, Marshall SW, Harding HP Jr, Guskiewicz KM. Nine-year risk of depression diagnosis increases with increasing self-reported concussions in retired professional football players. Am J Sports Med. 2012 Oct;40(10):2206-12. doi: 10.1177/0363546512456193. Epub 2012 Aug 24. PMID 22922518
- [Background] Clark MD, Varangis EML, Champagne AA, Giovanello KS, Shi F, Kerr ZY, Smith JK, Guskiewicz KM. Effects of Career Duration, Concussion History, and Playing Position on White Matter Microstructure and Functional Neural Recruitment in Former College and Professional Football Athletes. Radiology. 2018 Mar;286(3):967-977. doi: 10.1148/radiol.2017170539. Epub 2017 Oct 31. PMID 29087238
- [Background] Meehan WP 3rd, Taylor AM, Berkner P, Sandstrom NJ, Peluso MW, Kurtz MM, Pascual-Leone A, Mannix R. Division III Collision Sports Are Not Associated with Neurobehavioral Quality of Life. J Neurotrauma. 2016 Jan 15;33(2):254-9. doi: 10.1089/neu.2015.3930. Epub 2015 Jul 20. PMID 26193380
- [Background] Mannix R, Meehan WP 3rd, Pascual-Leone A. Sports-related concussions - media, science and policy. Nat Rev Neurol. 2016 Aug;12(8):486-90. doi: 10.1038/nrneurol.2016.99. Epub 2016 Jul 1. PMID 27364748
- [Background] Carson A. Concussion, dementia and CTE: are we getting it very wrong? J Neurol Neurosurg Psychiatry. 2017 Jun;88(6):462-464. doi: 10.1136/jnnp-2016-315510. Epub 2017 Apr 10. No abstract available. PMID 28396360
- [Background] Meehan W 3rd, Mannix R, Zafonte R, Pascual-Leone A. Chronic traumatic encephalopathy and athletes. Neurology. 2015 Oct 27;85(17):1504-11. doi: 10.1212/WNL.0000000000001893. Epub 2015 Aug 7. PMID 26253448
- [Background] Deshpande SK, Hasegawa RB, Rabinowitz AR, Whyte J, Roan CL, Tabatabaei A, Baiocchi M, Karlawish JH, Master CL, Small DS. Association of Playing High School Football With Cognition and Mental Health Later in Life. JAMA Neurol. 2017 Aug 1;74(8):909-918. doi: 10.1001/jamaneurol.2017.1317. PMID 28672325
- [Background] Baugh CM, Kroshus E, Kiernan PT, Mendel D, Meehan WP 3rd. Football Players' Perceptions of Future Risk of Concussion and Concussion-Related Health Outcomes. J Neurotrauma. 2017 Feb 15;34(4):790-797. doi: 10.1089/neu.2016.4585. Epub 2016 Sep 16. PMID 27526721
- [Background] Zemlan FP, Jauch EC, Mulchahey JJ, Gabbita SP, Rosenberg WS, Speciale SG, Zuccarello M. C-tau biomarker of neuronal damage in severe brain injured patients: association with elevated intracranial pressure and clinical outcome. Brain Res. 2002 Aug 23;947(1):131-9. doi: 10.1016/s0006-8993(02)02920-7. PMID 12144861
- [Background] Van Essen DC, Smith SM, Barch DM, Behrens TE, Yacoub E, Ugurbil K; WU-Minn HCP Consortium. The WU-Minn Human Connectome Project: an overview. Neuroimage. 2013 Oct 15;80:62-79. doi: 10.1016/j.neuroimage.2013.05.041. Epub 2013 May 16. PMID 23684880
- [Background] Smith SM, Beckmann CF, Andersson J, Auerbach EJ, Bijsterbosch J, Douaud G, Duff E, Feinberg DA, Griffanti L, Harms MP, Kelly M, Laumann T, Miller KL, Moeller S, Petersen S, Power J, Salimi-Khorshidi G, Snyder AZ, Vu AT, Woolrich MW, Xu J, Yacoub E, Ugurbil K, Van Essen DC, Glasser MF; WU-Minn HCP Consortium. Resting-state fMRI in the Human Connectome Project. Neuroimage. 2013 Oct 15;80:144-68. doi: 10.1016/j.neuroimage.2013.05.039. Epub 2013 May 20. PMID 23702415
- [Background] Glasser MF, Sotiropoulos SN, Wilson JA, Coalson TS, Fischl B, Andersson JL, Xu J, Jbabdi S, Webster M, Polimeni JR, Van Essen DC, Jenkinson M; WU-Minn HCP Consortium. The minimal preprocessing pipelines for the Human Connectome Project. Neuroimage. 2013 Oct 15;80:105-24. doi: 10.1016/j.neuroimage.2013.04.127. Epub 2013 May 11. PMID 23668970
- [Background] Hampshire A, MacDonald A, Owen AM. Hypoconnectivity and hyperfrontality in retired American football players. Sci Rep. 2013 Oct 17;3:2972. doi: 10.1038/srep02972. PMID 24135857
- [Background] Kaushal M, Espana LY, Nencka AS, Wang Y, Nelson LD, McCrea MA, Meier TB. Resting-state functional connectivity after concussion is associated with clinical recovery. Hum Brain Mapp. 2019 Mar;40(4):1211-1220. doi: 10.1002/hbm.24440. Epub 2018 Nov 19. PMID 30451340